CLINICAL TRIAL: NCT05383625
Title: Quadrivalent and Bivalent Human Papilloma Virus Vaccines in the Treatment of Common Recalcitrant Warts
Brief Title: Gardasil Versus Cervarix in the Treatment of Warts
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Hagar Nofal, Clinical Professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZU-IRB#5859/15-1-2020
Record Dates: First submitted 2022-05-12; First posted 2022-05-20 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Verruca Viral
MeSH Terms: interventions — Vaccines, Synthetic; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Quadrivalent vaccine (Experimental): Patient receive 0.1 ml of quadrivalent HPV vaccine intralesional every two weeks
  Interventions: Drug: Quadrivalent Human Papillomavirus (Types 6,11,16,18) Recombinant Vaccine
- Bivalent Vaccine (Experimental): Patient received 0.1 ml of bivalent HPV vaccine intralesional once every two weeks
  Interventions: Drug: Bivalent Human Papilloma Virus Vaccine
- Saline control (Placebo Comparator): Patient received 0.1 ml of intralesional saline once every two weeks
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Quadrivalent Human Papillomavirus (Types 6,11,16,18) Recombinant Vaccine — intralesional 0.1 ml every two weeks
  Arms: Quadrivalent vaccine
Drug: Bivalent Human Papilloma Virus Vaccine — Intralesional 0.1 ml every two weeks
  Arms: Bivalent Vaccine
Drug: Saline — intralesional into the largest warts every two weeks
  Arms: Saline control

SUMMARY:
Warts are common, benign, epidermal proliferations caused by HPV infecting skin and mucous membranes. Treatment of warts poses a true challenge despite existing variable therapeutic modalities, whether destructive or immunotherapeutic. Human papilloma virus (HPV) vaccines are FDA approved for the prevention of genital warts and wart related precancerous and cancerous lesions but they are not indicated for treatment of preexisting warts yet

DETAILED DESCRIPTION:
Approximately 35% of viral warts tend to be recalcitrant either showing no response to treatment or having prompt recurrences after treatment, causing frustration for both patients and physicians. Success rates vary significantly across patients and across different therapeutic interventions ranging from 7% to 90%.

Immunotherapy is proposed to enhance virus recognition by the cell mediated immunity, which allows the clearance of both treated and untreated warts and helps to prevent recurrences through induction of a long-term acquired immunity to HPV.

Few reports suggest the possibility of using quadrivalent or bivalent HPV vaccines as therapeutic modality rather than only preventive modality. This is a randomized controlled study to assess the efficacy and safety of quadrivalent and bivalent HPV vaccines in the treatment of warts

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients with recalcitrant multiple warts of any type. Warts were considered recalcitrant if they persisted for at least 6 months without any response to 2 different therapeutic modalities or more.
* Immunocompetent patients.
* Patients who do not receive any treatment of warts for at least 1 month before the start of study.

  * Patients who are able to understand and follow the study protocol and approve to sign the informed consent

Exclusion Criteria:

* Patients with acute febrile illness.
* Past history of asthma.
* Allergic skin disorders, such as generalized eczema, or severe urticaria.
* Pregnancy or lactation

  * History of hypersensitivity to the treatment vaccines.
  * Children
  * Immunocompromised patients
  * Patients unable to follow the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Therapeutic response | Through study completion for a maximum of 12 weeks, evaluation held at two weeks interval and at the end of treatment sessions (12th week visit)
  The percentage of patients in each group achieving complete, partial or no response at the end of the treatment sessions

SECONDARY OUTCOMES:
Safety measure | Through study completion every treatment session held at two weeks interval for a maximum of 5 sessions
  Immediate adverse events recorded by the treating physician within 1 hour post injection
Safety measure | Through study completion for a maximum of 12 weeks held every two weeks till the end of the treatment sessions (12th week visit)
  Delayed adverse events reported by the patients in between sessions
Recurrence | 6 months following the end of treatment sessions
  Percentage of patients experiencing recurrences in each group

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology department, Zagazig University Hospitals, Faculty of Medicine, Zagazig University, Zagazig, Select Region, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Nofal A, Marei A, Amer A, Amen H. Significance of interferon gamma in the prediction of successful therapy of common warts by intralesional injection of Candida antigen. Int J Dermatol. 2017 Oct;56(10):1003-1009. doi: 10.1111/ijd.13709. Epub 2017 Aug 8. PMID 28791682
- [Background] Nofal A, Marei A, Ibrahim AM, Nofal E, Nabil M. Intralesional versus intramuscular bivalent human papillomavirus vaccine in the treatment of recalcitrant common warts. J Am Acad Dermatol. 2020 Jan;82(1):94-100. doi: 10.1016/j.jaad.2019.07.070. Epub 2019 Jul 29. PMID 31369771
- [Background] Nofal A, Nofal E, Yosef A, Nofal H. Treatment of recalcitrant warts with intralesional measles, mumps, and rubella vaccine: a promising approach. Int J Dermatol. 2015 Jun;54(6):667-71. doi: 10.1111/ijd.12480. Epub 2014 Jul 29. PMID 25070525
- [Background] Landis MN, Lookingbill DP, Sluzevich JC. Recalcitrant plantar warts treated with recombinant quadrivalent human papillomavirus vaccine. J Am Acad Dermatol. 2012 Aug;67(2):e73-4. doi: 10.1016/j.jaad.2011.08.022. No abstract available. PMID 22794819
- [Background] Kreuter A, Waterboer T, Wieland U. Regression of cutaneous warts in a patient with WILD syndrome following recombinant quadrivalent human papillomavirus vaccination. Arch Dermatol. 2010 Oct;146(10):1196-7. doi: 10.1001/archdermatol.2010.290. No abstract available. PMID 20956677